CLINICAL TRIAL: NCT05303779
Title: Exercise Interventions of Eye Muscles for Improving Eye Control Post Strabismus Surgery
Brief Title: Exercise Interventions for Improving Eye Control Post Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Refaat Mohamed Abdel Wahid, principle investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003505
Record Dates: First submitted 2022-02-26; First posted 2022-03-31 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus | interventions — Dosage Forms; Eyeglasses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): experimental group will receive eye exercises in addition to medication and eye glasses post strabismus surgery
  Interventions: Other: Exercise Interventions of Eye Muscles; Drug: Medication and eye glasses
- control group (Active Comparator): control group will receive medication and eye glasses post strabismus surgery
  Interventions: Drug: Medication and eye glasses

INTERVENTIONS:
Other: Exercise Interventions of Eye Muscles — Application of eye exercise for improving eye control post strabismus surgery
  Other Names: experimental
  Arms: experimental group
Drug: Medication and eye glasses — medication and eye glasses used post strabismus surgery
  Other Names: control

SUMMARY:
The purpose of this study will be focused on the following issue:

1. The aim of this study is to determine therapeutic effect of postoperative eye exercises on improving eye control after the strabismus surgery.

HYPOTHESES:

It will be hypothesized that:

• Eye exercises have a positive effect on improving eye control post strabismus surgery.

RESEARCH QUESTION:"

• Do postoperative eye exercises improve eye control post strabismus surgery?

DETAILED DESCRIPTION:
Therapeutic procedures:

* Patient will be informed about measurement and treatment procedure before beginning of the treatment.
* Patient will be asked to follow physician instructions.
* Patients will be asked to avoid participation in any rehabilitation program prior to the study which may affect the result of the study.
* Measurement procedures will be applied for each patient.
* They will start the treatment program after 2 weeks of the surgery.

The subjects will be divided into two groups (experimental group and control group) with equal numbers of patients in each group:

Control group Participants within the control group will receive traditional care and medication following strabismus surgery.

Experimental group Participants within the experimental group will receive physiotherapy exercises beside traditional care and medication after strabismus surgery. Physical therapy exercises will apply in the office and home. Office exercises will involve palming exercise, pencil push-ups, brock string exercise, thumb exercise (Near-distance jump), balance board exercise, Proprioceptors Neuromuscular Facilitating (PNF) exercise, occlusive therapy, eye hand coordination and computer therapy. Office exercises will be done two sessions per week for three months. Each session will be about 1 hour. Exercises will also perform at home from the first session including eye exercises in all directions, pencil push-ups, thumb exercise (Near-distance jump),brock string exercise, and dominant eye occlusion for 1 hour daily.

ELIGIBILITY:
Inclusion Criteria:

* Criteria of selecting the patients include the following:
* Patients are both males and females.
* Their age will range from (5-15) years.
* Patients received strabismus operation.
* They will be selected from Outpatient Clinic of Research Institute of Ophthalmology.
* Patients will begin the training program after 2 weeks of operation.
* All types of strabismus surgery will be included.

Exclusion Criteria:

The subjects will be excluded from the study if they meet one of the following criteria;

* Muscular disorders that will impair performance during training.
* Any organic lesion in the eye.
* Neurological disorders.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.
* Children who can't understand the therapist's instructions and orders.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
changing in eye control | before the treatment and after 12 weeks (at the end of the treatment period )
  The level of control will be evaluated in each patient at both distance and near fixation using Intermittent Exotropia Control Scale.
  Fixation targets will be at 3 meters for distance fixation and it will be at 33 centimeters for near fixation.
  Intermittent Exotropia Control Scale
  5 = Constant exotropia 4 = Exotropia > 50% of the exam before dissociation 3 = Exotropia < 50% of the exam before dissociation 2 = No exotropia unless dissociated, recovers in > 5 seconds
  1 = No exotropia unless dissociated, recovers in 1-5 seconds 0 = No exotropia unless dissociated, recovers in < 1 second (phoria)
  The scale ranges from 0 (phoria, best control) to 5 (constant exotropia, worst control).

CONTACTS AND LOCATIONS:
Overall Officials: Amany Abdel Wahid, PhD, Principal Investigator — Lecturer
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No